CLINICAL TRIAL: NCT04491877
Title: Safety, Immunogenicity, Infectivity, and Dose-Finding Study of an Investigational Live-Attenuated Respiratory Syncytial Virus (RSV) Vaccine in Infants and Toddlers
Brief Title: Study of an Live-Attenuated Respiratory Syncytial Virus Vaccine in Infants and Toddlers
Acronym: VAD00001
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAD00001; U1111-1238-1869 (Registry Identifier: ICTRP)
Record Dates: First submitted 2020-07-27; First posted 2020-07-29 (Actual); Results first posted 2024-06-13 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Respiratory Syncytial Virus Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study was performed in an observer-blind fashion. Investigators and study staff who conducted the safety assessment and the participants did not know which vaccine is administered. Only the study staff who prepare and administer the vaccine and were not involved with the safety evaluation knew which vaccine was administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Cohort 1 (RSV vaccine formulation 1) (Experimental): 1 administration of RSV vaccine formulation 1 on Day 0
  Interventions: Biological: RSV vaccine formulation 1
- Cohort 1 (Placebo) (Placebo Comparator): 1 administration of placebo on Day 0
  Interventions: Biological: Placebo
- Cohort 2 (RSV vaccine formulation 1) (Experimental): 2 administrations of RSV vaccine formulation 1 on Day 0 and Day 56
  Interventions: Biological: RSV vaccine formulation 1
- Cohort 2 (Placebo) (Placebo Comparator): 2 administrations of placebo on Day 0 and Day 56
  Interventions: Biological: Placebo
- Cohort 3 (RSV vaccine formulation 2) (Experimental): 1 administration of RSV vaccine formulation 2 on Day 0
  Interventions: Biological: RSV vaccine formulation 2
- Cohort 3 (Placebo) (Placebo Comparator): 1 administration of placebo on Day 0
  Interventions: Biological: Placebo
- Cohort 4 (RSV vaccine formulation 1) (Experimental): 2 administrations of RSV vaccine formulation 1 on Day 0 and Day 56
  Interventions: Biological: RSV vaccine formulation 1
- Cohort 4 (RSV vaccine formulation 2) (Experimental): 2 administrations of RSV vaccine formulation 2 on Day 0 and Day 56
  Interventions: Biological: RSV vaccine formulation 2
- Cohort 4 (Placebo) (Placebo Comparator): 2 administrations of placebo on Day 0 and Day 56
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: RSV vaccine formulation 1 — Pharmaceutical form: Suspension of virus Route of administration: Intranasal
  Arms: Cohort 1 (RSV vaccine formulation 1); Cohort 2 (RSV vaccine formulation 1); Cohort 4 (RSV vaccine formulation 1)
Biological: RSV vaccine formulation 2 — Pharmaceutical form: Suspension of virus Route of administration: Intranasal
  Arms: Cohort 3 (RSV vaccine formulation 2); Cohort 4 (RSV vaccine formulation 2)
Biological: Placebo — Pharmaceutical form: Suspension Route of administration: Intranasal
  Arms: Cohort 1 (Placebo); Cohort 2 (Placebo); Cohort 3 (Placebo); Cohort 4 (Placebo)

SUMMARY:
The primary objectives of the study were:

* To assess the safety profile of each dose of the study product after each and any administration in all infants and toddlers regardless of baseline serostatus.
* To characterize the Respiratory Syncytial Virus (RSV) A serum neutralizing antibody responses to the study product in each vaccine group after vaccination in RSV-naïve participants.

The secondary objectives of the study were:

* To quantify the amount of vaccine virus shed by each participant by baseline serostatus.
* To determine the proportion of vaccinated infants and toddlers in each vaccine group infected with the vaccine virus at D56 (56 days after vaccination 1) for Cohorts 1, 2, 3 and 4, and at Day 84 (28 days after vaccination 2) for Cohorts 2 and 4 by baseline serostatus.
* To characterize the RSV A serum neutralizing antibody responses to the study product in each vaccine group after vaccination in RSV-experienced participants.
* To characterize serum RSV anti-F immunoglobulin G (IgG) antibody responses to the study product in each vaccine group after vaccination by baseline serostatus.
* To characterize serum RSV antibody responses (RSV A-neutralizing and anti-RSV F IgG) to the study product in each vaccine group after the RSV surveillance season or at least 5 months after the last vaccine administration by baseline serostatus.

DETAILED DESCRIPTION:
Study duration per participant was maximum 12 months

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria :

* Aged 6 through 18 months at Day 0.
* Informed consent form has been signed and dated by the parent(s) or other legally acceptable representative (and by independent witness if required by local regulations).
* Participant and parent / guardian / legally acceptable representative are able to attend all scheduled visits and to comply with all trial procedures

Exclusion Criteria:

* Born at less than 34 weeks gestation
* Born at less than 37 weeks gestation and less than 1 year of age at the time
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Probable or confirmed case of Coronavirus Disease 2019 (COVID-19).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the trial or to a vaccine containing any of the same substances
* Any chronic illness

  • Chronic illness may include, but is not limited to, cardiac disorders, lung disease (including any history of reactive airway disease, receipt of bronchodilator therapy, or medically diagnosed wheezing), renal disorders, auto-immune disorders, diabetes, psychomotor diseases, and known congenital or genetic diseases
* Any history of medically diagnosed wheezing
* Any acute febrile, respiratory or gastrointestinal illness in the past 24 hours that according to investigator judgment is significant enough to interfere with successful inoculation on the day of vaccination. A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided
* Any previous anaphylactic reaction
* Current suspected or documented developmental disorder, delay, or other developmental problem
* Receipt of any of the following vaccines prior to enrollment:

  * any influenza vaccine within 7 days prior, or
  * any inactivated vaccine or live-attenuated rotavirus vaccine within the 14 days prior, or
  * any live vaccine, other than rotavirus vaccine, within the 28 days prior, or
  * another investigational vaccine or investigational drug within 28 days prior
* Previous receipt of a licensed or investigational RSV vaccine or previous receipt or planned administration of any anti-RSV product (such as ribavirin or RSV immune immune globulins [IG] or RSV monoclonal antibody)
* Receipt of immune globulins, blood or blood-derived products in the past 6 months prior to enrolment
* Receipt of any of the following medications within 3 days prior to study enrollment (Day 0):

  * systemic antibacterial, antiviral, antifungal, anti-parasitic, or antituberculous agents, whether for treatment or prophylaxis, or
  * intranasal medications, or
  * other prescription medication except as permitted concomitant medications (prescription or non-prescription) including nutritional supplements, medications for gastroesophageal reflux, eye drops, and topical medications, including (but not limited to) cutaneous (topical) steroids, topical antibiotics, and topical antifungal agents
* Receipt of salicylate (aspirin) or salicylate-containing products within the 28 days prior to enrollment (Day 0)
* Any previous vaccine-associated adverse reaction that was Grade 3 or above. Note: if grading is not possible, determine if the reaction was considered severe or life threatening; if so, it is exclusionary.
* Scheduled administration of the following after planned inoculation:

  * any influenza vaccine within 7 days after, or
  * inactivated vaccine or live-attenuated rotavirus vaccine within the 14 days after, or
  * any live vaccine other than rotavirus in the 28 days after, or
  * another investigational vaccine or investigational drug in the 56 days after.
* Any previous receipt of supplemental oxygen therapy in a home or hospital setting, except the temporary receipt of supplemental oxygen for transient tachypnea in newborn
* Member of a household that contains an immunocompromised individual, including, but not limited to:

  * a person who is HIV infected
  * a person who has received chemotherapy within the 12 months prior to enrollment
  * a person receiving immunosuppressant agents
  * a person living with a solid organ or bone marrow transplant
* Participation at the time of study enrollment (or in the 6 weeks preceding the first trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Member of a household that contains, or will contain, an infant who is less than 6 months of age at the enrollment date (or in the 6 weeks preceding the first trial vaccination) through Day 28
* Member of a household that contains another child/other children who is/are, or is/are scheduled to be, enrolled in this study in the same year AND the date of enrollment will not be concurrent with the other participant(s) living in the household (i.e., all eligible children from the same household must be enrolled on the same date)
* Attends a daycare facility and shares a daycare room with infants less than 6 months of age, and parent/guardian is unable or unwilling to suspend daycare for 28 days following inoculation
* Deprived of freedom in an emergency setting or hospitalized involuntarily
* Identified as a natural or adopted child of the Investigator or employee with direct involvement in the proposed study

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 259 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2023-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (29):
- United States (25):
  - Matrix Clinical Research-Site Number:8400012, Gardena, California
  - Paradigm Clinical Research-Site Number:8400026, La Mesa, California
  - Matrix Clinical Research-Site Number:8400032, Los Angeles, California
  - California Research Foundation-Site Number:8400016, San Diego, California
  - Elite Clinical Trials, Inc.-Site Number:8400001, Blackfoot, Idaho
  - Leavitt Clinical Research-Site Number:8400036, Idaho Falls, Idaho
  - Snake River Research-Site Number:8400022, Idaho Falls, Idaho
  - The South Bend Clinic Center for Research-Site Number:8400024, South Bend, Indiana
  - Alliance for Multispeciality Research-Site Number:8400014, El Dorado, Kansas
  - AMR - Newton-Site Number:8400002, Newton, Kansas
  - Michael W. Simon, MD, PSC-Site Number:8400013, Lexington, Kentucky
  - Benchmark Research-Site Number:8400006, Covington, Louisiana
  - Nola Research Works-Site Number:8400017, New Orleans, Louisiana
  - Clinical Research Institute-Site Number:8400053, Minneapolis, Minnesota
  - Boeson Research-Site Number:8400011, Missoula, Montana
  - Be Well Clinical Studies-Site Number:8400054, Lincoln, Nebraska
  - Meridian Clinical Research - Norfolk-Site Number:8400005, Norfolk, Nebraska
  - MedPharmics Inc-Site Number:8400040, Albuquerque, New Mexico
  - East Carolina University/Brody Medical Sciences Building-Site Number:8400043, Greenville, North Carolina
  - Coastal Pediatric Research-Site Number:8400031, Charleston, South Carolina
  - Tribe Clinical Research-Site Number:8400027, Greenville, South Carolina
  - FMC Science-Site Number:8400042, Lampasas, Texas
  - JBR Clinical Research-Site Number:8400041, Salt Lake City, Utah
  - Pediatric Associates of Charlottesville North-Site Number:8400007, Charlottesville, Virginia
  - National Clinical Research Inc-Site Number:8400004, Richmond, Virginia
- Chile (2):
  - Investigational Site Number :1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number :1520004, Santiago, Reg Metropolitana de Santiago
- Honduras (2):
  - Investigational Site Number :3400001, San Pedro Sula
  - Investigational Site Number :3400002, Tegucigalpa

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Idoko OT, Vargas SL, Bueso A, Rivera D, Edward H, Simon M, Banooni P, Berger S, Janicot S, Vercasson C, Pallardy S, Nteene R, Adhikarla H, Gerchman E, Gasparotto M, Gallichan S, Rivas E, Buchholz UJ, Collins PL, Sesay S, Gurunathan S, De Bruijn I, Dhingra MS. Live-Attenuated Intranasal RSV Vaccine in Infants and Toddlers. NEJM Evid. 2025 Sep;4(9):EVIDoa2500026. doi: 10.1056/EVIDoa2500026. Epub 2025 Aug 26. PMID 40856556
- See also: VAD00001 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25364&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 26 centers in the United States, Chile and Honduras between 17 September 2020 and 13 April 2023.
Pre-assignment Details: A total of 259 participants were enrolled and randomized in the study.
Groups:
- Cohort 1: Respiratory Syncytial Virus (RSV) Low Dose: Participants received a single low dose intranasal spray of RSV ΔNS2/Δ1313/I1314L vaccine (RSVt) on Day 0.
- Cohort 1: Placebo; Cohort 3: Placebo: Participants received a single intranasal spray of placebo on Day 0.
- Cohort 2: RSV Low Dose; Cohort 4: RSV Low Dose: Participants received low dose RSVt intranasal spray once daily on Days 0 and 56.
- Cohort 2: Placebo; Cohort 4: Placebo: Participants received placebo intranasal spray once daily on Days 0 and 56.
- Cohort 3: RSV High Dose: Participants received a single high dose intranasal spray of RSVt on Day 0.
- Cohort 4: RSV High Dose: Participants received high dose RSVt intranasal spray once daily on Days 0 and 56.
Period: Overall Study
Arm/Group | Cohort 1: Respiratory Syncytial Virus (RSV) Low Dose | Cohort 1: Placebo | Cohort 2: RSV Low Dose | Cohort 2: Placebo | Cohort 3: RSV High Dose | Cohort 3: Placebo | Cohort 4: RSV Low Dose | Cohort 4: RSV High Dose | Cohort 4: Placebo
Started | 18 | 18 | 11 | 10 | 10 | 12 | 61 | 58 | 61
Completed | 17 | 16 | 9 | 8 | 10 | 10 | 56 | 51 | 57
Not Completed | 1 | 2 | 2 | 2 | 0 | 2 | 5 | 7 | 4
Not completed — Protocol Deviation | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Parent/Guardian | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 5 | 3
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Randomized participants included all participants allocated to a vaccine group.
Groups:
- Cohort 1: RSV Low Dose: Participants received a single low dose intranasal spray of RSVt on Day 0.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: RSV Low Dose | Cohort 1: Placebo | Cohort 2: RSV Low Dose | Cohort 2: Placebo | Cohort 3: RSV High Dose | Cohort 3: Placebo | Cohort 4: RSV Low Dose | Cohort 4: RSV High Dose | Cohort 4: Placebo | Total
Number analyzed (Participants) | 18 | 18 | 11 | 10 | 10 | 12 | 61 | 58 | 61 | 259
Age, Continuous [Mean (Standard Deviation); unit: months] | 11.2 (4.51) | 11.8 (3.09) | 11.4 (4.01) | 10.8 (4.13) | 12.1 (3.11) | 12.8 (3.95) | 10.4 (3.17) | 10.6 (3.63) | 10.6 (3.78) | 10.9 (3.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 4 | 5 | 4 | 3 | 31 | 25 | 32 | 123
  Male | 10 | 7 | 7 | 5 | 6 | 9 | 30 | 33 | 29 | 136
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 11 | 9 | 30
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 0 | 0 | 2 | 1 | 3 | 1 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  White | 16 | 16 | 11 | 10 | 10 | 10 | 41 | 35 | 38 | 187
  Mixed Origin | 1 | 0 | 0 | 0 | 0 | 0 | 8 | 9 | 13 | 31
  Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Immediate Unsolicited Systemic Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant or in a clinical investigation participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. An unsolicited AE is an observed AE that does not fulfill the conditions pre-listed in the case report book (CRB) in terms of diagnosis and/or onset window post-vaccination. Systemic AEs are all AEs that were not injection or administration site reactions. Immediate events are recorded to capture medically relevant unsolicited systemic AEs (including those related to the product administered) that occur within the first 30 minutes after vaccination.
Time Frame: Cohorts 1 and 3: Within 30 minutes after vaccination on Day 0; Cohorts 2 and 4: Within 30 minutes after vaccination on Days 0 and 56
Population: The Safety analysis set (SafAS) included participants who received at least 1 administration of the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: RSV Low Dose | Cohort 1: Placebo | Cohort 2: RSV Low Dose | Cohort 2: Placebo | Cohort 3: RSV High Dose | Cohort 3: Placebo | Cohort 4: RSV Low Dose | Cohort 4: RSV High Dose | Cohort 4: Placebo
Number analyzed (Participants) | 17 | 18 | 10 | 10 | 10 | 12 | 61 | 57 | 61
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

2. Primary Outcome: Number of Participants With Solicited Administration Site and Systemic Reactions
Description: All noxious and unintended responses to a medicinal product related to any dose are considered adverse reactions (AR). A solicited reaction is an "expected" AR (sign or symptom) observed and reported under the conditions (nature and onset) pre-listed in the protocol and CRB. An administration site reaction is an AR at and around the administration site. Systemic ARs are all ARs that are not injection or administration site reactions.
Time Frame: Cohorts 1 and 3: Within 28 days after vaccination on Day 0; Cohorts 2 and 4: Within 28 days after vaccination on Days 0 and 56
Population: The SafAS included participants who received at least 1 administration of the study vaccine. Only participants with available data are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: RSV Low Dose | Cohort 1: Placebo | Cohort 2: RSV Low Dose | Cohort 2: Placebo | Cohort 3: RSV High Dose | Cohort 3: Placebo | Cohort 4: RSV Low Dose | Cohort 4: RSV High Dose | Cohort 4: Placebo
Number analyzed (Participants) | 17 | 18 | 10 | 10 | 10 | 11 | 59 | 56 | 61
Participants
  Solicited administration site reactions | 15 | 12 | 8 | 7 | 9 | 6 | 53 | 44 | 53
  Solicited systemic reactions | 14 | 16 | 9 | 9 | 9 | 9 | 50 | 46 | 51

3. Primary Outcome: Number of Participants With Unsolicited Adverse Events
Description: An AE is any untoward medical occurrence in a participant or in a clinical investigation participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. An unsolicited AE is an observed AE that does not fulfill the conditions pre-listed in the CRB in terms of diagnosis and/or onset window post-vaccination.
Time Frame: as for outcome 2
Population: The SafAS included participants who received at least 1 administration of the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: RSV Low Dose | Cohort 1: Placebo | Cohort 2: RSV Low Dose | Cohort 2: Placebo | Cohort 3: RSV High Dose | Cohort 3: Placebo | Cohort 4: RSV Low Dose | Cohort 4: RSV High Dose | Cohort 4: Placebo
Number analyzed (Participants) | 17 | 18 | 10 | 10 | 10 | 12 | 61 | 57 | 61
Participants | 6 | 2 | 2 | 5 | 0 | 2 | 43 | 35 | 46

4. Primary Outcome: Number of Participants With Adverse Events of Special Interest (AESIs)
Description: An AESI is one of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor can be appropriate.
Time Frame: as for outcome 2
Population: The SafAS included participants who received at least 1 administration of the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: RSV Low Dose | Cohort 1: Placebo | Cohort 2: RSV Low Dose | Cohort 2: Placebo | Cohort 3: RSV High Dose | Cohort 3: Placebo | Cohort 4: RSV Low Dose | Cohort 4: RSV High Dose | Cohort 4: Placebo
Number analyzed (Participants) | 17 | 18 | 10 | 10 | 10 | 12 | 61 | 57 | 61
Participants | 3 | 0 | 0 | 0 | 0 | 1 | 20 | 11 | 20

5. Primary Outcome: Number of Participants With Medically Attended Adverse Events (MAAEs)
Description: An MAAE is a new onset or a worsening of a condition that prompts the participant or participant's parent/guardian/legally authorized representative to seek unplanned medical advice at a physician's office or Emergency Department.
Time Frame: as for outcome 2
Population: The SafAS included participants who received at least 1 administration of the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: RSV Low Dose | Cohort 1: Placebo | Cohort 2: RSV Low Dose | Cohort 2: Placebo | Cohort 3: RSV High Dose | Cohort 3: Placebo | Cohort 4: RSV Low Dose | Cohort 4: RSV High Dose | Cohort 4: Placebo
Number analyzed (Participants) | 17 | 18 | 10 | 10 | 10 | 12 | 61 | 57 | 61
Participants | 3 | 1 | 0 | 4 | 0 | 1 | 36 | 29 | 36

6. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An SAE is any untoward medical occurrence that at any dose results in death or is life-threatening or requires inpatient hospitalization or prolongation of existing hospitalization or results in persistent or significant disability/incapacity or is a congenital anomaly/birth defect or is an important medical event.
Time Frame: From the first study vaccine administration (Day 0) up to end of the study, maximum of 12 months
Population: The SafAS included participants who received at least 1 administration of the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: RSV Low Dose | Cohort 1: Placebo | Cohort 2: RSV Low Dose | Cohort 2: Placebo | Cohort 3: RSV High Dose | Cohort 3: Placebo | Cohort 4: RSV Low Dose | Cohort 4: RSV High Dose | Cohort 4: Placebo
Number analyzed (Participants) | 17 | 18 | 10 | 10 | 10 | 12 | 61 | 57 | 61
Participants | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 2

7. Primary Outcome: Geometric Mean Titers Against RSV A Neutralizing Antibody in RSV-Naïve Participants
Description: RSV A neutralizing antibody measured by microneutralization. RSV-naïve participants are defined as undetectable serum anti-RSV A IgA antibodies.
Time Frame: Cohorts 1 and 3: Day 56; Cohorts 2 and 4: Days 56 and 84
Population: The full analysis set (FAS) included all randomized participants who received at least 1 administration of the study vaccine. Only participants analyzed at each specific time point are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1: RSV Low Dose | Cohort 1: Placebo | Cohort 2: RSV Low Dose | Cohort 2: Placebo | Cohort 3: RSV High Dose | Cohort 3: Placebo | Cohort 4: RSV Low Dose | Cohort 4: RSV High Dose | Cohort 4: Placebo
Number analyzed (Participants) | 11 | 9 | 6 | 8 | 7 | 9 | 29 | 22 | 29
titer
  Day 56 | 75.9 [39.7 to 145] | 32.8 [22.0 to 48.7] | 180 [55.4 to 585] | 27.5 [21.7 to 35.0] | 99.2 [40.9 to 241] | 17.9 [11.4 to 27.9] | 83.7 [49.5 to 142] | 79.4 [47.2 to 134] | 20.6 [16.4 to 25.9]
  Day 84: number analyzed (Participants) | 0 | 0 | 6 | 8 | 0 | 0 | 28 | 21 | 27
  Day 84 |  |  | 181 [65.2 to 500] | 19.8 [12.1 to 32.1] |  |  | 142 [86.4 to 232] | 107 [70.0 to 163] | 26.3 [18.8 to 37.0]

8. Secondary Outcome: Titer of Vaccine Virus Shedding Measured by Reverse Transcription Polymerase Chain Reaction (RT-PCR)
Description: Shedding of the attenuated RSV vaccine strain in nasal swab samples was evaluated by RSV quantitative RT-PCR (qRT-PCR) assay, which specifically detected and quantified RSVt ΔNS2 vaccine strain (RSV ΔNS2/Δ1313/I1314L) in human nasal swab samples.
Time Frame: Cohorts 1 and 3: Day 7; Cohorts 2 and 4: Days 7 and 63
Population: The SafAS included participants who received at least 1 administration of the study vaccine.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Cohort 1: RSV Low Dose | Cohort 1: Placebo | Cohort 2: RSV Low Dose | Cohort 2: Placebo | Cohort 3: RSV High Dose | Cohort 3: Placebo | Cohort 4: RSV Low Dose | Cohort 4: RSV High Dose | Cohort 4: Placebo
Number analyzed (Participants) | 7 | 0 | 10 | 0 | 7 | 0 | 23 | 20 | 0
log10 copies/mL
  After first vaccination | 5.02 (1.03) |  | 6.27 (0.883) |  | 5.82 (0.666) |  | 5.16 (0.940) | 5.21 (0.985) |
  After second vaccination: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 3 | 0
  After second vaccination |  |  | 5.35 (NA) — Standard deviation was not calculable because only one participant was analyzed. |  |  |  | 5.10 (1.78) | 5.76 (1.21) |

9. Secondary Outcome: Percentage of Participants Infected With Vaccine Virus at Days 56 and 84
Description: Infection is defined as detection of vaccine virus in nasal swab by RT-PCR and/or a >= 4-fold rise in RSV A serum neutralizing antibody titers, or in RSV serum anti-F immunoglobulin G (IgG) antibody titers.
Time Frame: Cohorts 1 and 3: Day 56; Cohorts 2 and 4: Days 56 and 84
Population: The FAS included all randomized participants who received at least 1 administration of the study vaccine. Only participants analyzed at each specific time point are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: RSV Low Dose | Cohort 1: Placebo | Cohort 2: RSV Low Dose | Cohort 2: Placebo | Cohort 3: RSV High Dose | Cohort 3: Placebo | Cohort 4: RSV Low Dose | Cohort 4: RSV High Dose | Cohort 4: Placebo
Number analyzed (Participants) | 17 | 16 | 10 | 8 | 10 | 10 | 49 | 48 | 50
percentage of participants
  After first vaccination | 82.4 [56.6 to 96.2] | 12.5 [1.6 to 38.3] | 100 [69.2 to 100] | 0 [0 to 36.9] | 100 [69.2 to 100] | 0 [0 to 30.8] | 63.3 [48.3 to 76.6] | 58.3 [43.2 to 72.4] | 4.0 [0.5 to 13.7]
  After second vaccination: number analyzed (Participants) | 0 | 0 | 7 | 7 | 0 | 0 | 39 | 41 | 48
  After second vaccination |  |  | 71.4 [29.0 to 96.3] | 0 [0 to 41.0] |  |  | 64.1 [47.2 to 78.8] | 51.2 [35.1 to 67.1] | 18.8 [8.9 to 32.6]

10. Secondary Outcome: Geometric Mean Titers Against RSV A Neutralizing Antibody in RSV-Experienced Participants
Description: RSV A neutralizing antibody measured by microneutralization. RSV-experienced participants are defined as detectable serum anti-RSV A IgA antibodies. CI= confidence interval.
Time Frame: Cohorts 1 and 3: Day 56; Cohorts 2 and 4: Days 56 and 84
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1: RSV Low Dose | Cohort 1: Placebo | Cohort 2: RSV Low Dose | Cohort 2: Placebo | Cohort 3: RSV High Dose | Cohort 3: Placebo | Cohort 4: RSV Low Dose | Cohort 4: RSV High Dose | Cohort 4: Placebo
Number analyzed (Participants) | 6 | 7 | 1 | 0 | 2 | 1 | 14 | 20 | 23
titer
  Day 56: number analyzed (Participants) | 6 | 7 | 1 | 0 | 2 | 1 | 14 | 20 | 22
  Day 56 | 134 [37.6 to 476] | 52.1 [22.7 to 120] | 672 [NA to NA] — 95% CI was not calculable when number of participants with available data for the considered endpoint (e.g., number of analyzed participants) were <= 5 or STD = 0 |  | 409 [NA to NA] — 95% CI was not calculable when number of participants with available data for the considered endpoint (e.g., number of analyzed participants) were <= 5 or STD = 0 | 15.0 [NA to NA] — 95% CI was not calculable when number of participants with available data for the considered endpoint (e.g., number of analyzed participants) were <= 5 or STD = 0 | 120 [60.8 to 238] | 96.0 [65.0 to 142] | 73.5 [44.0 to 123]
  Day 84: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 14 | 20 | 23
  Day 84 |  |  | 243 [NA to NA] — 95% CI was not calculable when number of participants with available data for the considered endpoint (e.g., number of analyzed participants) were <= 5 or STD = 0 |  |  |  | 120 [65.1 to 221] | 102 [70.5 to 148] | 96.7 [44.9 to 208]

11. Secondary Outcome: Geometric Mean Titers Against Serum Anti-F Immunoglobulin G (IgG) Antibody
Description: The IgG antibodies to RSV F antigen was measured using the anti RSV F IgG ELISA. RSV-naïve and RSV-experienced participants are defined as undetectable or detectable serum anti-RSV A IgA antibodies, respectively.
Time Frame: Cohorts 1 and 3: Day 56; Cohorts 2 and 4: Days 56 and 84
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1: RSV Low Dose | Cohort 1: Placebo | Cohort 2: RSV Low Dose | Cohort 2: Placebo | Cohort 3: RSV High Dose | Cohort 3: Placebo | Cohort 4: RSV Low Dose | Cohort 4: RSV High Dose | Cohort 4: Placebo
Number analyzed (Participants) | 11 | 9 | 6 | 8 | 7 | 9 | 27 | 21 | 29
titer
  RSV-naïve participants: Day 56 | 32.8 [18.1 to 59.6] | 15.0 [6.77 to 33.4] | 58.8 [18.0 to 191] | 8.63 [6.20 to 12.0] | 48.7 [26.3 to 90.0] | 7.50 [NA to NA] — 95% CI was not calculable when number of participants with available data for the considered endpoint (e.g., number of analyzed participants) were <= 5 or STD = 0 | 43.2 [27.1 to 69.1] | 45.6 [28.1 to 73.9] | 10.4 [7.70 to 14.1]
  RSV-naïve participants: Day 84: number analyzed (Participants) | 0 | 0 | 6 | 8 | 0 | 0 | 26 | 20 | 26
  RSV-naïve participants: Day 84 |  |  | 135 [55.5 to 331] | 8.72 [6.11 to 12.4] |  |  | 93.1 [49.0 to 177] | 61.8 [35.1 to 109] | 12.5 [8.30 to 18.7]
  RSV-experienced participants: Day 56: number analyzed (Participants) | 6 | 7 | 1 | 0 | 2 | 1 | 14 | 20 | 21
  RSV-experienced participants: Day 56 | 205 [29.5 to 1421] | 38.5 [7.60 to 195] | 230 [NA to NA] — 95% CI was not calculable when number of participants with available data for the considered endpoint (e.g., number of analyzed participants) were <= 5 or STD = 0 |  | 337 [NA to NA] — 95% CI was not calculable when number of participants with available data for the considered endpoint (e.g., number of analyzed participants) were <= 5 or STD = 0 | 7.50 [NA to NA] — 95% CI was not calculable when number of participants with available data for the considered endpoint (e.g., number of analyzed participants) were <= 5 or STD = 0 | 215 [93.8 to 491] | 251 [139 to 455] | 124 [50.7 to 304]
  RSV-experienced participants: Day 84: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 14 | 19 | 23
  RSV-experienced participants: Day 84 |  |  | 165 [NA to NA] — 95% CI was not calculable when number of participants with available data for the considered endpoint (e.g., number of analyzed participants) were <= 5 or STD = 0 |  |  |  | 250 [108 to 576] | 287 [175 to 473] | 221 [76.8 to 635]

12. Secondary Outcome: Geometric Mean Titers Against RSV A Neutralizing Antibody After the RSV Surveillance Season
Description: RSV A neutralizing antibody measured by microneutralization. RSV-naïve and RSV-experienced participants are defined as undetectable or detectable serum anti-RSV A IgA antibodies, respectively.
Time Frame: Cohorts 1 and 3: Within 5 months after vaccination on Day 0; Cohorts 2 and 4: Within 5 months after vaccination on Day 56
Population: The FAS included all randomized participants who received at least 1 administration of the study vaccine. Only participants analyzed for this outcome measure are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1: RSV Low Dose | Cohort 1: Placebo | Cohort 2: RSV Low Dose | Cohort 2: Placebo | Cohort 3: RSV High Dose | Cohort 3: Placebo | Cohort 4: RSV Low Dose | Cohort 4: RSV High Dose | Cohort 4: Placebo
Number analyzed (Participants) | 17 | 15 | 6 | 7 | 9 | 9 | 37 | 40 | 47
titer | 73.2 [45.5 to 118] | 24.4 [16.2 to 36.5] | 303 [119 to 768] | 16.6 [13.0 to 21.3] | 294 [125 to 691] | 108 [32.4 to 362] | 112 [69.3 to 180] | 123 [71.7 to 211] | 56.6 [33.2 to 96.5]

13. Secondary Outcome: Geometric Mean Titers Against Serum Anti-F Immunoglobulin G Antibody After the RSV Surveillance Season
Description: as for outcome 11
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1: RSV Low Dose | Cohort 1: Placebo | Cohort 2: RSV Low Dose | Cohort 2: Placebo | Cohort 3: RSV High Dose | Cohort 3: Placebo | Cohort 4: RSV Low Dose | Cohort 4: RSV High Dose | Cohort 4: Placebo
Number analyzed (Participants) | 16 | 15 | 6 | 7 | 8 | 8 | 36 | 39 | 44
titer | 63.7 [28.7 to 141] | 14.2 [7.51 to 27.0] | 388 [95.2 to 1581] | 8.63 [6.12 to 12.2] | 296 [92.6 to 948] | 272 [35.8 to 2067] | 222 [124 to 397] | 300 [159 to 568] | 94.4 [43.6 to 204]

ADVERSE EVENTS:
Time Frame: From the first study vaccine administration (Day 0) up to end of the study, maximum of 12 months
Description: Analysis was performed on the safety analysis set.
Arm/Group | Cohort 1: RSV Low Dose | Cohort 1: Placebo | Cohort 2: RSV Low Dose | Cohort 2: Placebo | Cohort 3: RSV High Dose | Cohort 3: Placebo | Cohort 4: RSV Low Dose | Cohort 4: RSV High Dose | Cohort 4: Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/18 | 0/10 | 0/10 | 0/10 | 0/12 | 0/61 | 0/57 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/18 | 1/10 | 0/10 | 0/10 | 1/12 | 2/61 | 1/57 | 2/61
Other Adverse Events (participants affected / at risk) | 15/17 | 17/18 | 10/10 | 9/10 | 9/10 | 10/12 | 55/61 | 49/57 | 59/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: RSV Low Dose (N=17) | Cohort 1: Placebo (N=18) | Cohort 2: RSV Low Dose (N=10) | Cohort 2: Placebo (N=10) | Cohort 3: RSV High Dose (N=10) | Cohort 3: Placebo (N=12) | Cohort 4: RSV Low Dose (N=61) | Cohort 4: RSV High Dose (N=57) | Cohort 4: Placebo (N=61)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intussusception (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atypical Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Syncytial Virus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchial Obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulite (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: RSV Low Dose (N=17) | Cohort 1: Placebo (N=18) | Cohort 2: RSV Low Dose (N=10) | Cohort 2: Placebo (N=10) | Cohort 3: RSV High Dose (N=10) | Cohort 3: Placebo (N=12) | Cohort 4: RSV Low Dose (N=61) | Cohort 4: RSV High Dose (N=57) | Cohort 4: Placebo (N=61)
Conjunctivitis Allergic (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 5 (5) | 6 (7)
Teething (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 3 (3) | 3 (5) | 4 (5) | 2 (2) | 1 (1) | 22 (29) | 23 (30) | 28 (30)
Crying (General disorders) | 9 (9) | 8 (8) | 7 (10) | 6 (9) | 7 (7) | 3 (3) | 31 (43) | 28 (41) | 29 (39)
Pyrexia (General disorders) | 1 (1) | 5 (5) | 1 (2) | 1 (1) | 1 (1) | 2 (2) | 21 (27) | 19 (20) | 22 (23)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 2 (2)
Ear Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Myringitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 19 (26) | 20 (22) | 18 (22)
Otitis Media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Otitis Media Acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 3 (3)
Sinusitis Bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 3 (3) | 4 (4)
Viral Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Animal Bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod Sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 6 (6) | 6 (6) | 6 (7) | 5 (6) | 7 (7) | 3 (3) | 29 (40) | 38 (50) | 33 (44)
Somnolence (Nervous system disorders) | 5 (5) | 5 (5) | 6 (8) | 5 (6) | 5 (5) | 4 (4) | 23 (31) | 30 (39) | 20 (24)
Irritability (Psychiatric disorders) | 13 (13) | 12 (12) | 8 (10) | 8 (10) | 7 (7) | 9 (9) | 40 (60) | 37 (53) | 38 (53)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 5 (5) | 5 (5)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 6 (6) | 7 (9) | 6 (9) | 7 (7) | 5 (5) | 46 (68) | 43 (68) | 51 (68)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 10 (10) | 8 (9) | 6 (9) | 8 (8) | 5 (5) | 52 (77) | 43 (70) | 47 (66)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2023-01-19): https://cdn.clinicaltrials.gov/large-docs/77/NCT04491877/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-30): https://cdn.clinicaltrials.gov/large-docs/77/NCT04491877/SAP_001.pdf